CLINICAL TRIAL: NCT02573012
Title: Prospective, Multicentre, Placebo-controlled, Double-blind Interventional Study to Compare the Efficacy of Maintenance Treatment With Tocilizumab With or Without Glucocorticoid Discontinuation in Rheumatoid Arthritis Patients
Brief Title: Study to Compare the Efficacy of Tocilizumab With or Without Glucocorticoid Discontinuation in Rheumatoid Arthritis Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MA29585; 2014-004673-16 (EudraCT Number)
Record Dates: First submitted 2015-10-01; First posted 2015-10-09 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Prednisone; tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Tocilizumab+prednisone (constant dose) (Experimental): Participants will receive tocilizumab at a dose of 162 milligram (mg) once a week subcutaneously; and prednisone at a dose of 5 milligram per day (mg/day) or matching placebo orally for 24 weeks.
  Interventions: Drug: Placebo matched to prednisone; Drug: Prednisone; Biological: Tocilizumab
- Tocilizumab+prednisone (tapering dose) (Experimental): Participants will receive tocilizumab at a dose of 162 milligram (mg) once a week subcutaneously; and prednisone at a dose of 5 milligram per day (mg/day) with 1 mg decrements every 4 weeks or matching placebo orally for 24 weeks.
  Interventions: Drug: Placebo matched to prednisone; Drug: Prednisone; Biological: Tocilizumab

INTERVENTIONS:
Drug: Placebo matched to prednisone — Participants will receive placebo matched to prednisone orally for 24 weeks.
Drug: Prednisone — Participants will receive prednisone either at a constant dose of 5 mg/day, or 5 mg/day with 1 mg decrements every 4 weeks orally for 24 weeks.
Biological: Tocilizumab — Participants will receive tocilizumab at a dose of 162 mg once a week subcutaneously for 24 weeks.

SUMMARY:
This Phase IIIb/IV, two-arm, randomized, double-blind, placebo-controlled, parallel-group, international, multicenter trial compares the change in disease activity (as assessed by Disease Activity Score in 28 joints [DAS28] erythrocyte sedimentation rate [ESR]) from randomization to Week 24 post-randomization, in participants with stable low disease activity [LDA] (DAS28 ESR score less than or equal to [<=] 3.2) who receive tocilizumab, and have been randomized to either continue or taper prednisone in a double-blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

Tocilizumab-experienced participants:

* Comply with the requirements of the study protocol (including treatment on an outpatient basis)
* Rheumatoid arthritis (RA) of greater than or equal to (>=) 6 months duration diagnosed according to the revised 1987 American College of Rheumatology (ACR) criteria or 2010 ACR / European League Against Rheumatism (EULAR) criteria
* Have received tocilizumab either subcutaneous (162 milligram [mg] once in a week) or intravenously (8 milligram per kilogram [mg/kg] once every 4 weeks) for the treatment of RA for at least 24 weeks prior to randomization
* Have received 5 - 15 milligrams per day [mg/day] of glucocorticoids (prednisone or equivalent) for the treatment of RA for at least 20 weeks prior to screening
* Currently receiving 5 mg/day of prednisone
* Have attained and maintained LDA (DAS28 ESR score <=3.2) or remission (DAS28 ESR score less than [<] 2.6) for at least 4 weeks prior to randomization

Tocilizumab-naïve participants:

* Comply with the requirements of the study protocol (including treatment on an outpatient basis)
* RA of >=6 months duration diagnosed according to the revised 1987 ACR criteria or 2010 ACR / EULAR criteria
* Have active RA (defined as DAS28 ESR score greater than [>] 3.2)
* Are considered by the investigator as inadequate responders to conventional synthetic disease-modifying anti-rheumatic drugs (csDMARDs) or biologic disease-modifying anti-rheumatic drugs (bDMARDs)
* Are receiving 5 - 15 mg/day prednisone (or equivalent) for the treatment of RA

Exclusion Criteria:

General

* Major surgery (including joint surgery) within 8 weeks prior to screening, or planned major surgery during the study and up to 6 months after randomization
* Pregnant women or nursing (breastfeeding) mothers
* In females of childbearing potential, a positive serum pregnancy test at screening
* Females of childbearing potential unwilling or unable to use a reliable means of contraception (for example, physical barrier [participant or partner], contraceptive pill or patch, spermicide and barrier, or intrauterine device) during study treatment and for a minimum of 3 months after the last dose of tocilizumab
* Body weight of >=150 kilogram (kg)
* Lack of peripheral venous access

Disease-related

* RA of functional Class 4, as defined by the ACR Classification of Functional Status in Rheumatoid Arthritis
* Rheumatic autoimmune disease other than RA, including systemic lupus erythematosus, mixed connective tissue disease, scleroderma, polymyositis, or significant systemic involvement secondary to RA (for example, vasculitis, pulmonary fibrosis, or Felty syndrome). Secondary Sjögren syndrome with RA may be allowed per the discretion of the investigator
* Diagnosed with juvenile idiopathic arthritis or juvenile RA and/or RA before the age of 16 years
* Prior or current inflammatory joint disease other than RA (for example, gout, Lyme disease, sero-negative spondyloarthropathy, including reactive arthritis, psoriatic arthritis, arthropathy of inflammatory bowel disease), or prior or current joint infections
* Previous history of primary or secondary adrenal insufficiency

Previous or Concomitant Prohibited Therapy

* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of screening
* Previous treatment with any cell-depleting therapies, including investigational agents or approved therapies (for example, CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19, anti-CD20)
* Treatment with intravenous gamma globulin, plasmapheresis or Prosorba column within 6 months of screening
* Intraarticular (IA) or parenteral glucocorticoids for the treatment of RA within 4 weeks prior to screening
* Previous treatment with glucocorticoids for conditions other than RA, at any dose and in any formulation used continuously for >1 week, during the last 1 year prior to screening. Topical glucocorticoid creams or ointments for the treatment of skin conditions (for example eczema) are allowed
* Immunization with a live/attenuated vaccine within 30 days prior to screening. Participants must agree not to take live attenuated vaccines (including seasonal nasal flu vaccine, varicella vaccine for shingles or chickenpox, vaccines for measles, mumps or rubella without or with varicella [MMR or MMRV], oral polio vaccine and vaccines for yellow fever), within 30 days before the Screening Visit, throughout the duration of the trial and for 60 days following the last dose of study drug
* Any previous treatment with alkylating agents such as chlorambucil or with total lymphoid irradiation

Laboratory Exclusion Criteria

* Inadequate haematological, renal and liver function
* Positive hepatitis B surface antigen or hepatitis C antibody Previous or Concomitant Conditions
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* Evidence of current serious uncontrolled cardiovascular (including uncontrolled hyperlipidemia), nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (including uncontrolled diabetes mellitus) or gastrointestinal (GI) disease
* Current liver disease as determined by the investigator
* History of diverticulitis, peptic ulcer disease, diverticulosis requiring antibiotic treatment, or chronic ulcerative lower GI disease such as Crohn's disease, ulcerative colitis, or other symptomatic lower gastrointestinal conditions that might predispose to perforations
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial, or other opportunistic infections (including, but not limited to, tuberculosis [TB] and atypical mycobacterial disease, hepatitis B and C, Epstein-Barr virus, cytomegalovirus and herpes zoster, but excluding fungal infections of nail beds)
* Neuropathies or other conditions that might interfere with pain evaluation unless related to primary disease under investigation
* Any major episode of infection requiring hospitalization or treatment with intravenous antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* Active TB requiring treatment within the previous 3 years (participants previously treated for TB with no recurrence within 3 years are permitted). All Track tocilizumab-naïve participants must be screened for latent TB and if positive, should be treated following local practice guidelines prior to initiating tocilizumab
* History of or currently active, primary or secondary immunodeficiency
* Evidence of active malignant disease, malignancies diagnosed within the previous 10 years (including haematological malignancies and solid tumours, except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that was excised and cured), or breast cancer diagnosed within the previous 20 years
* History of alcohol, drug or chemical abuse within 1 year prior to screening
* Pre-existing central nervous system (CNS) demyelination or seizure disorders
* Any medical or psychological condition that in the opinion of the principal investigator would interfere with safe completion of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (39):
- France (5):
  - Hopital Pellegrin; Rhumatologie, Bordeaux
  - Hopital de La Source, Orléans
  - Hopital Cochin; Rhumatologie B, Paris
  - Hopital Hautepierre; Rhumatologie, Strasbourg
  - Hopital Purpan; Rhumatologie, Toulouse
- Germany (20):
  - Praxis Dr. med. Reiner Kurthen, Aachen
  - Asklepios Kllinikum Bad Abbach; Klinik für Rheumatologie und Klinische Immunologie, Bad Abbach
  - Rheumatologische Gemeinschaftspraxis Grafschaft, Dr. med. Dorothea Pick, Dr. med. Christopher Amberg, Bad Neuenahr-Ahrweiler
  - Charité Campus Mitte, Med.Klinik, Rheumatologie und Klinische Immunologie, Berlin
  - SchlossPark-Klinik Berlin; Int. Med. II, Rheum. Osteo, Berlin
  - Klinik der Uni zu Köln; Klinik für Innere Medizin, Cologne
  - Rheumatologisches MVZ Dresden GmbH, Dres. Holger Schwenke, Reiner Schwenke, Annekatrin Georgi, Dresden
  - MVZ Ambulantes Rheumazentrum, Erfurt
  - Dres. Florian Schuch, Ruediger de la Camp, Martin Hammerschmidt u.w., Erlangen
  - Universitätsklinikum Hamburg-Eppendorf Zentrum f.Innere Medizin Med.Klinik III, Hamburg
  - Praxis Dr.med. Maria Höhle, Hamburg
  - Rheumapraxis PD Dr.med. Bernhard Heilig, Heidelberg
  - Rheumatologische Facharztpraxis Maren Sieburg, Magdeburg
  - SMO.MD GmbH, Zentrum für klinische Studien, Magdeburg
  - Klinikum der Universitat Munchen; Bereich Pettenkoferstr; Rheumaeinheit der medizinischen Klinik IV, München
  - Praxiszentrum St. Bonifatius, München
  - Rheumapraxis an der Hase, Osnabrück
  - Rheumazentrum Ratingen - Studienambulanz, Ratingen
  - Rheumatologische Schwerpunktpraxis am Feuersee, Stuttgart
  - Universitätsklinikum Würzburg; Medizinische Klinik und Poliklinik II; Rheumatologie/Immunologie, Würzburg
- Italy (3):
  - Arcispedale Santa Maria Nuova; Reumatologia, Reggio Emilia, Emilia-Romagna
  - Irccs Policlinico San Matteo; Reumatologia Adulti, Pavia, Lombardy
  - Ospedale Careggi Villa Monnatessa ; Sezione Di Reumatologia, Florence, Tuscany
- Russia (5):
  - FSBI Scientific Research Institute of Clinical and Experimental Lymphology of SB of RAMS, Novosibirsk
  - Perm Regional Clinical Hospital, Perm
  - SBEI of HPE "Northwestern State Medical University n.a. I.I.Mechnikov" of MoH of RF, Saint Petersburg
  - Republican clinical hospital named after G.G. Kuvatov, Ufa
  - City Clinical Hospital # 2, Vladivostok
- Serbia (5):
  - Institute of Rheumatology, Belgrade
  - Military Medical Academy; Clinic of Rheumatology, Belgrade
  - Institute of Rheumatology and Cardiovascular Diseases; Rheumatology, Niška Banja
  - Clinical Center of Vojvodina, Novi Sad
  - Special hospital for rheumatic diseases Novi Sad, Novi Sad
- Hopital Farhat Hached; Service Rhumatologie, Sousse, Tunisia

REFERENCES:
- [Derived] Burmester GR, Buttgereit F, Bernasconi C, Alvaro-Gracia JM, Castro N, Dougados M, Gabay C, van Laar JM, Nebesky JM, Pethoe-Schramm A, Salvarani C, Donath MY, John MR; SEMIRA collaborators. Continuing versus tapering glucocorticoids after achievement of low disease activity or remission in rheumatoid arthritis (SEMIRA): a double-blind, multicentre, randomised controlled trial. Lancet. 2020 Jul 25;396(10246):267-276. doi: 10.1016/S0140-6736(20)30636-X. PMID 32711802

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 314 participants were enrolled in the study; 55 participants discontinued the study prior to randomization; 259 participants were randomized.
Groups:
- Tocilizumab+Prednisone (Tapering Dose): Participants will receive tocilizumab at a dose of 162 milligram (mg) once a week subcutaneously or 8 mg/kg intravenously every 4 weeks; and prednisone at a dose of 5 milligram per day (mg/day) with 1 mg decrements every 4 weeks or matching placebo orally for 24 weeks.
- Tocilizumab+Prednisone (Constant Dose): Participants will receive tocilizumab at a dose of 162 milligram (mg) once a week subcutaneously or 8 mg/kg intravenously every 4 weeks; and prednisone at a dose of 5 milligram per day (mg/day) or matching placebo orally for 24 weeks.
Period: Overall Study
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Started | 131 | 128
Completed | 116 | 113
Not Completed | 15 | 15
Not completed — Adverse Event | 5 | 5
Not completed — Lack of Efficacy | 5 | 4
Not completed — Non-compliance | 1 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Study Ended per Protocol | 1 | 0
Not completed — Physician Decision | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose) | Total
Number analyzed (Participants) | 131 | 128 | 259
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (14.0) | 54.0 (12.8) | 54.4 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 97 | 200
  Male | 28 | 31 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 120 | 114 | 234
  Unknown or Not Reported | 10 | 14 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 0 | 0 | 0
  White | 129 | 123 | 252
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score in 28 Joints - Erythrocyte Sedimentation Rate (DAS28-ESR) at Week 24 Post-randomization
Description: The DAS28 is a combined index for measuring disease activity in rheumatic arthritis (RA) and includes swollen and tender joint count, erythrocyte sedimentation rate (ESR), and general health (GH) status. The index is calculated with the following formula: DAS28 = (0.56 × √(TJC28)) + (0.28 × √(SJC28)) + (0.7 × log(ESR)) + (0.014 × GH), where TJC28 = tender joint count and SJC28 = swollen joint count, each on 28 joints. GH = a patient's global assessment of disease activity in the previous 24 hours on a 100-millimeter (mm) visual analog scale (left end = no disease activity [symptom-free and no arthritis symptoms], right end = maximum disease activity [maximum arthritis disease activity]). When ESR equaled 0 mm/hr, it was set to 1 mm/hr. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. A positive change in score indicates worsening, and a negative change indicates improvement.
Time Frame: Baseline to Week 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
Score on a scale | 0.538 [0.346 to 0.729] | -0.075 [-0.271 to 0.121]
Statistical Analysis 1: Comparison: Tocilizumab+Prednisone (Tapering Dose) vs Tocilizumab+Prednisone (Constant Dose); Test type: Superiority; p = 0.001, ANCOVA; Least Square Means = 0.613, 95% CI 2-sided [0.346 to 0.879]

2. Secondary Outcome: Treatment Success
Description: Treatment success was defined as the percentage of participants with stable low disease activity (LDA) (DAS28-ESR score ≤ 3.2) at Week 24 post-randomization, who did not suffer a flare due to RA and who showed no confirmed adrenal insufficiency that required replacement therapy. DAS28 has the following standardized cut-offs for disease activity and remission: DAS28 > 5.1 = high disease activity; DAS28 between 3.2 and 5.1 = moderate disease activity; DAS28 ≤ 3.2 = low disease activity; DAS28 ≤ 2.6 = remission.
Time Frame: Week 24
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
Percentage of Participants | 64.9 [56.1 to 73.0] | 77.3 [69.1 to 84.3]
Statistical Analysis 1: Comparison: Tocilizumab+Prednisone (Tapering Dose) vs Tocilizumab+Prednisone (Constant Dose); Test type: Superiority; p = 0.018, Regression, Logistic; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.285 to 0.889]
Statistical Analysis 2: Comparison: Tocilizumab+Prednisone (Tapering Dose) vs Tocilizumab+Prednisone (Constant Dose); Test type: Superiority; p = 0.021, Cochran-Mantel-Haenszel; Relative Risk = 0.833, 95% CI 2-sided [0.714 to 0.972]

3. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Week 24
Description: Clinical Disease Activity Index (CDAI) is an index for measuring disease activity in rheumatoid arthritis (RA). The index is calculated using the following formula: CDAI = number of swollen joints using the 28-joint count (SJC28) + number of tender joints using the 28-joint count (TJC28) + patient global assessment of disease (PGA) based on 10 centimeter (cm) visual analog scale (VAS) + physician global assessment of disease (PhGA) based on 10 cm VAS. VAS assessments involved a 100 mm horizontal scale from 0 (no disease activity) to 10 (maximum disease activity). Total CDAI scores range from 0 to 76, with higher scores indicating increased disease activity. A positive change in score indicates worsening, and a negative change indicates improvement.
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
Score on a scale | 2.663 [1.454 to 3.872] | 0.321 [-0.914 to 1.556]
Statistical Analysis 1: Comparison: Tocilizumab+Prednisone (Tapering Dose) vs Tocilizumab+Prednisone (Constant Dose); Test type: Superiority; p = 0.006, ANCOVA; Least Square Mean = 2.342, 95% CI 2-sided [0.661 to 4.023]

4. Secondary Outcome: Percentage of Participants With >=1 Flare
Description: Percentage of participants with >=1 flare
Time Frame: 24 weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
Percentage of Participants | 26.0 | 10.9

5. Secondary Outcome: Time to First RA Flare
Description: The mean time of onset for the first RA flare since randomization.
Time Frame: Randomization to 24 weeks
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
Weeks | 15.64 (7.13) | 12.11 (7.96)

6. Secondary Outcome: Percentage of Visits With RA Flares
Time Frame: Randomization to 24 weeks
Measure: Number; unit: Percentage of visits with flares
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
Percentage of visits with flares
  1 Visit | 16.0 | 7.0
  2 Visits | 6.9 | 3.9
  3 Visits | 2.3 | 0
  >3 Visits | 0.8 | 0

7. Secondary Outcome: Percentage of Participants With >=1 Administration of Flare Rescue Medication
Description: The proportion of participants with at least one administration of RA flare rescue medication.
Time Frame: Randomization to 24 weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
Percentage of Participants | 20.6 | 6.3

8. Secondary Outcome: Time to First Administration of Flare Rescue Medication
Description: Time of onset of first administration of RA flare rescue medication since randomization date
Time Frame: Randomization to 24 weeks
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
Weeks | 13.59 (6.77) | 8.76 (5.26)

9. Secondary Outcome: Number of Administrations of Flare Rescue Medication
Description: Proportion of participants who received courses of RA flare rescue medication by number of courses received.
Time Frame: Randomization to 24 weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
Percentage of Participants
  0 courses | 79.4 | 93.8
  1 course | 15.3 | 3.9
  2 courses | 4.6 | 1.6
  3 courses | 0 | 0.8
  >3 courses | 0.8 | 0

10. Secondary Outcome: Cumulative Prednisone Exposure (Dose)
Description: In Post-randomization prednisone arm, Cumulative dose = (number of capsules taken during week 1 to 4 * 1 mg) + (3/4 * number of capsules taken during week 5 to 8 * 1 mg) + (1/2 * number of capsules taken during week 9 to 12 * 1 mg) + (1/4 * number of capsules taken during week 13 to 16 * 1 mg). In continued arm, cumulative dose = (1/4 * number of capsule taken * 5 mg).
  Cumulative prednisone dose is defined as cumulative blinded prednisone + cumulative flare rescue prednisone.
Time Frame: Randomization to 24 weeks
Population: Safety Population. The cumulative flare rescue prednisone dose population is based upon the number of participants who required rescue treatment.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
mg
  Cumulative blinded prednisone dose: number analyzed (Participants) | 131 | 127
  Cumulative blinded prednisone dose | 267.099 (40.048) | 769.459 (175.882)
  Cumulative flare rescue prednisone dose: number analyzed (Participants) | 27 | 8
  Cumulative flare rescue prednisone dose | 98.519 (51.921) | 121.875 (54.898)
  Cumulative prednisone dose: number analyzed (Participants) | 131 | 127
  Cumulative prednisone dose | 287.405 (63.184) | 777.136 (172.881)

11. Secondary Outcome: Percentage of Participants Who Maintain LDA (DAS28 ESR Score <=3.2) or Remission (DAS28 ESR Score <2.6) and the Percentage of Participants Who Maintain the Baseline Disease Activity Level
Description: The proportion of participants who maintained LDA and the proportion of participants who maintained the baseline disease activity level at Week 24.
  LDA was defined as DAS28 ESR score <= 3.2. Remission was defined as DAS28 ESR score <= 2.6. Participants who maintained the baseline activity was defined as DAS28-ESR at Week 24 <= DAS28-ESR at baseline.
Time Frame: Randomization to Week 24
Population: Intent to Treat population. The number of participants for LDA at Week 24 and Remission at Week 24 are based upon the number with LDA at baseline and DAS28-ESR ≤ 2.6 at baseline respectively.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
Percentage of Participants
  LDA at baseline: number analyzed (Participants) | 128 | 124
  LDA at baseline | 97.7 | 96.9
  LDA at Week 24: number analyzed (Participants) | 128 | 124
  LDA at Week 24 | 73.4 | 83.1
  Baseline DAS28-ESR ≤ 2.6: number analyzed (Participants) | 103 | 98
  Baseline DAS28-ESR ≤ 2.6 | 78.6 | 76.6
  Remission at Week 24: number analyzed (Participants) | 103 | 98
  Remission at Week 24 | 61.2 | 81.6
  Maintained baseline activity at Week 24 | 36.6 | 54.7

12. Secondary Outcome: Percentage of Participants Who Permanently Discontinue Study Treatment Due to Insufficient Flare Control
Description: Percentage of participants who permanently discontinue study treatment due to insufficient flare control
Time Frame: 24 weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
Percentage of Participants | 0 | 0.8

13. Secondary Outcome: Changes From Baseline in American College of Rheumatology (ACR) Core Set Components at Week 24: Swollen 66 Joint Counts
Description: Count of swollen joints based upon 66 assessed joints.
Time Frame: Baseline to Week 24
Measure: Mean (Standard Deviation); unit: Swollen joints
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
Swollen joints | 0.129 (6.687) | -0.107 (1.618)

14. Secondary Outcome: Changes From Baseline in American College of Rheumatology (ACR) Core Set Components at Week 24: Tender 68 Joint Counts
Description: Count of tender joints based on 68 assessed joints.
Time Frame: Baseline to Week 24
Measure: Mean (Standard Deviation); unit: Tender joints
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
Tender joints | 0.793 (7.764) | -0.330 (2.729)

15. Secondary Outcome: Changes From Baseline in American College of Rheumatology (ACR) Core Set Components at Week 24: Patient's Assessment of Pain
Description: The ACR patient's assessment of pain is scored on a visual analog scale (VAS) from 0 (no pain) to 100 mm (unbearable pain). A positive change in score indicates worsening, and a negative change indicates improvement.
Time Frame: Baseline to Week 24
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
mm | 4.648 (24.315) | -8.010 (25.980)

16. Secondary Outcome: Changes From Baseline in American College of Rheumatology (ACR) Core Set Components at Week 24: Patient's Global Assessment of Disease Activity
Description: The ACR patient's global assessment of disease activity is scored on a visual analog scale (VAS) from 0 (symptom-free and no arthritis symptoms) to 100 mm (maximum arthritis disease activity). A positive change in score indicates worsening, and a negative change indicates improvement.
Time Frame: Baseline to Week 24
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
cm | 0.280 (2.000) | -0.153 (1.506)

17. Secondary Outcome: Changes From Baseline in American College of Rheumatology (ACR) Core Set Components at Week 24: Physician's Global Assessment of Disease Activity
Description: The ACR physician's global assessment of disease activity is scored on a visual analog scale (VAS) from 0 (symptom-free and no arthritis symptoms) to 100 mm (maximum arthritis disease activity). A positive change in score indicates worsening, and a negative change indicates improvement.
Time Frame: Baseline to Week 24
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
cm | 0.345 (1.463) | -0.248 (1.167)

18. Secondary Outcome: Changes From Baseline in American College of Rheumatology (ACR) Core Set Components at Week 24: Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: A measure of self-perceived disability containing 20 questions in eight categories and including additional section about aid from other people and devices needed to correct the disabilities. Scores range from 0 to 3, with higher scores indicating worse disability.
Time Frame: Baseline to Week 24
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
Score on a scale | 0.167 (0.486) | -0.087 (0.527)

19. Secondary Outcome: Changes From Baseline in American College of Rheumatology (ACR) Core Set Components at Week 24: High Sensitivity C-Reactive Protein (hsCRP)
Description: Change from baseline in the acute phase reactant hsCRP
Time Frame: Baseline to Week 24
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
mg/dL | -0.135 (1.470) | -0.040 (0.277)

20. Secondary Outcome: Changes From Baseline in American College of Rheumatology (ACR) Core Set Components at Week 24: Erythrocyte Sedimentation Rate (ESR)
Description: Change from baseline in the acute phase reactant ESR
Time Frame: Baseline to Week 24
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
mm/hr | 1.517 (7.892) | -0.679 (5.433)

21. Secondary Outcome: Changes From Baseline in Rheumatoid Arthritis Impact of Disease (RAID) Final Score
Description: The RAID is a participant-completed questionnaire specific for RA consisting of a 0-10 rating for pain, functional disability, fatigue, sleep, physical well-being, emotional well-being and coping. Scores are weighted to produce a final numerical result. A positive change in score indicates worsening, and a negative change indicates improvement.
Time Frame: Baseline and Week 24
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
Score on a scale | 0.469 (2.109) | -0.220 (1.940)

22. Secondary Outcome: Changes From Baseline in Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP) Score
Description: The WPAI:SHP is a 6-item questionnaire to measure performance impairment of work and regular daily activity and yields 4 types of scores: work time missed (absenteeism), impairment while working (presenteeism or reduced on-the-job effectiveness), overall work impairment (WI) (work productivity loss or absenteeism plus presenteeism) and activity impairment (daily activity impairment). Total score and each score range from 0 (not affected/no impairment) to 100 (completely affected/impaired). Higher scores indicate greater impairment and less productivity. A positive change in score indicates impairment, and a negative change indicates improvement.
Time Frame: Baseline and Week 24
Population: Intent to Treat population.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
Score on a scale
  Percent work time missed due to problem: number analyzed (Participants) | 38 | 34
  Percent work time missed due to problem | 4.535 (23.283) | 0.572 (31.455)
  Percent impairment while working due to problem: number analyzed (Participants) | 47 | 41
  Percent impairment while working due to problem | -0.851 (24.920) | -5.584 (23.343)
  Percent overall work impairment due to problem: number analyzed (Participants) | 36 | 32
  Percent overall work impairment due to problem | 6.219 (29.223) | -6.191 (30.531)
  Percent activity impairment due to problem: number analyzed (Participants) | 103 | 105
  Percent activity impairment due to problem | 3.398 (23.786) | -4.190 (21.608)

23. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) at Week 24
Description: The SDAI is the numerical sum of 5 outcome parameters: tender and swollen joint count based on a 28-joint assessment, patient and physician global assessment of disease activity according to 100-mm visual analog scale (VAS) and level of C-reactive protein in milligrams per deciliter (mg/dL, normal <1 mg/dl). The total SDAI score range is 0-86, where higher scores indicate increased disease activity. A positive change in score indicates worsening, and a negative change indicates improvement.
Time Frame: Randomization to Week 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
Number analyzed (Participants) | 131 | 128
Score on a scale | 2.511 [1.296 to 3.727] | 0.248 [-0.994 to 1.489]
Statistical Analysis 1: Comparison: Tocilizumab+Prednisone (Tapering Dose) vs Tocilizumab+Prednisone (Constant Dose); Test type: Superiority; p = 0.009, ANCOVA; Least Square Means = 2.264, 95% CI [0.574 to 3.953]

ADVERSE EVENTS:
Time Frame: Randomization to Week 28
Arm/Group | Tocilizumab+Prednisone (Tapering Dose) | Tocilizumab+Prednisone (Constant Dose)
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/128
Serious Adverse Events (participants affected / at risk) | 7/131 | 4/128
Other Adverse Events (participants affected / at risk) | 46/131 | 21/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab+Prednisone (Tapering Dose) (N=131) | Tocilizumab+Prednisone (Constant Dose) (N=128)
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 1
CELLULITIS GANGRENOUS (Infections and infestations) | 0 | 1
BLOOD GLUCOSE FLUCTUATION (Investigations) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
SCIATICA (Nervous system disorders) | 0 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 1
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab+Prednisone (Tapering Dose) (N=131) | Tocilizumab+Prednisone (Constant Dose) (N=128)
NASOPHARYNGITIS (Infections and infestations) | 13 | 9
DIARRHOEA (Gastrointestinal disorders) | 7 | 5
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 9 | 3
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 9 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT02573012/Prot_SAP_000.pdf